CLINICAL TRIAL: NCT05898035
Title: Postoperative Symptoms Following Endodontic Microsurgery Performed by Piezoelectric Osteotomy Versus Conventional Osteotomy: A Randomized Clinical Trial
Brief Title: Postoperative Symptoms Following Endodontic Microsurgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Lama Awawdeh, Professor, King Abdullah University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KingAbdullahUH
Record Dates: First submitted 2023-03-02; First posted 2023-06-12 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Pain Postoperative; Swelling Lips & Face
Keywords: Microsurgery, Pain, swelling, Piezo surgery
MeSH Terms: conditions — Pain, Postoperative; Facies; Pain

STUDY DESIGN:
Intervention Model Description: This a randomized prospective clinical study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezo endodontic surgery (Experimental): The osteotomy will be applied under magnification with a surgical operating microscope (at the apical third of the root .Osteotomy will be done with the Piezosurgery touch
  Interventions: Procedure: Endodontic Microsurgery
- Conventional endodontic surgery (Active Comparator): The osteotomy will be applied under magnification with a surgical operating microscope at the apical third of the root .Osteotomy will be done with air motor high speed hand-piece and round bur with copious irrigation
  Interventions: Procedure: Endodontic Microsurgery

INTERVENTIONS:
Procedure: Endodontic Microsurgery — Osteotomy will be done either with air motor high speed hand-piece and round bur with copious irrigation or with Piezosurgery touch. After the soft tissue curettage and uncovering the root apex , the last 3 mm of the root apex will be resected perpendicular to the long axis of the tooth at ( 0 - 10) degree bevel , using either conventional dental hand-piece or piezotome (Piezotome Cube by ACTEON ).The resected root will be rinsed , dried and and stained with 1% methylene blue dye after which , it will be inspected carefully under high magnification, to identify possible reasons for the non surgical root canal treatment failure. Subsequently, ultrasonic apical preparation will be performed. After achieving adequate haemostasis with Epinephrine pellets. Biodentine®retrograde filling material will be placed. The flap will be re-approximated and interrupted suture using non-absorbable monofilament size 5-0 suture will be applied. Finally, Post-operative parallel Digital view.

SUMMARY:
Aims: The purpose of this randomized clinical trial is to assess and compare the post operative pain, swelling and quality of life after endodontic microsurgery using either conventional osteotomy or piezoelectric osteotomy . The PICO question that will be used is Does endodontic microsurgery using piezoelectric osteotomy have similar clinical performance in terms of post operative pain and swelling to that of endodontic microsurgery using conventional hand-piece osteotomy.

Material and methods:

based on solid inclusion criteria , a total of 44 patients in need of endodontic microsurgery will be randomly distributed into two groups (n=22) according to the osteotomy technique: conventional and piezoelectric osteotomy. A standardized microsurgical technique will be employed. After the microsurgery procedure, a pain questionnaire that contain visual analogue scale will be given to each patient to evaluate the pain incidence and intensity at 5 time intervals, 24 hours, 48 hours, 72 hours, 96 hours and 120 hours. The patients will be recalled as well, at days 2 and 7 to evaluate the swelling. Statistical analysis will be performed using chi-square test and linear regression analysis.

DETAILED DESCRIPTION:
This randomized prospective clinical study will be conducted at the postgraduate clinics, Department of Conservative Dentistry, at Jordan University of Science and Technology.

Ethical approval will be sought from the JUST Institutional ethics and human Research Board (IRB) committee.

Sample size and randomization A total of 44 adult patients will be recruited for this clinical trial. Participants will be randomly allocated to one of the two treatment modalities. Randomization will be carried out by sealed envelope online software.

For the observational part of the study, no randomization or blinding will be applied. Patients will be treated free of charge and their travel expenses will be compensated for all follow up visits.

Preoperative management :

Clinical and radiographic assessment :

- The patient demographic information, chief complaint and history of the chief complaint, medical and dental history will be registered. A thorough extra-oral and intra-oral examination will be undertaken (an existing swelling , sinus tracts, quality of coronal restoration margins and its history, occlusal relations, gingival biotype , any gingival recession and periodontal assessment ) will be registered .

Percussion and palpating tests will be applied. Pre-operative parallel Digital view will be obtained using film holder showing the entire lesion and at least 2 mm beyond it. Limited view cone beam computed tomography scan of the diseased tooth will be obtained for each patient preoperatively (SFV).

Root length and axis, Lesion size and features, bone crest level and any radiographic abnormality will be interpreted and registered.

All patients will receive periodontal scaling a week or two before the surgery. Surgical procedure Prior to surgery , patients will be asked to rinse their mouth with chlorhexidine 0.12% . After which, local anesthesia containing epinephrine will be given. The surgical flap design and procedure will be selected as per case deem , and the flap will be elevated gently and retracted.

The Root apex will be located and osteotomy will be applied. The resected root will be rinsed , dried and and stained with 1% methylene blue dye after which , it will be inspected carefully under high magnification, to identify possible reasons for the non surgical root canal treatment failure. Subsequently, ultrasonic apical preparation will be performed. After achieving adequate haemostasis with Epinephrine pellets (Gingi-Pak , California state , USA),Biodentine retrograde filling material will be placed. The flap will be re-approximated and interrupted suture using non-absorbable monofilament size 5-0 suture will be applied. Finally, Post-operative parallel Digital view will be obtained using film holder showing the entire lesion and at least 2 mm beyond it.

Post-operative management :

Immediately after the microsurgery the patients will be asked to apply cold ice packs on the surgical site for 20 mins at the clinic, during this time the post-operative instructions will be given .

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers .
* Teeth that are periodontally healthy.
* Age (18-65)

Exclusion Criteria:

* Patients with an active systematic diseases that may affect the outcome
* Medically compromised patients on long term medications.
* Patients who had received analgesics or antibiotics prior to surgery will be postponed.
* Cases where orthograde endodontic treatment is feasible
* Teeth with poor prognosis.
* Teeth with an active periodontal disease (pocket depth > 5 mm).
* Emotionally distressed patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
changes in pain severity | to measure changes in the pain severity at 3 hours, 24 hours , 48 hours , 72 hours and 120 hours.
  visual analogue scale that is calibrated between (no discomfort ) and end with (very server pain ),
Swelling size changes | At the second and seventh days after the microsurgery, patients will be re-called for the determination of edema and swelling
  Changes in amount of swelling will be measured by measuring distance between fixed points in patient face.

CONTACTS AND LOCATIONS:
Overall Officials: Lama A Awawdeh, PhD, Principal Investigator — Jordan University of Science and Technolgoy
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No